CLINICAL TRIAL: NCT01264172
Title: Identification of the Cutaneous and Muscular Microcirculation and Inflammatory Response After Minimal-invasive Osteosynthesis of the Proximal Femur
Brief Title: Identification of Microcirculation and Inflammation After Minimal-invasive Osteosynthesis of the Proximal Femur
Acronym: MicroProxFem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC-A10-28
Record Dates: First submitted 2010-12-19; First posted 2010-12-21 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Level of Pain
Keywords: Functional outcome; Microcirculation; Inflammatory response
MeSH Terms: interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PCCP, Proximal femur fracture (Active Comparator): Patients, who received a minimal-invasive surgical treatment with the PCCP-plate
  Interventions: Procedure: PCCP
- Osteosythesis with nails, prox. femur frac. (Active Comparator): Patients, who received a minimal-invasive surgical treatment including a osteosynthesis with nails
  Interventions: Procedure: Osteosynthesis with nails
- DHS, proximal femur fracture (Active Comparator): Patients, who received a conventional surgical treatment with the dynamic hip screw (DHS)
  Interventions: Procedure: DHS

INTERVENTIONS:
Procedure: PCCP — PCCP: an minimal-invasive surgery technique, in wich a special plate is pushed in position and fixed through 2 small approaches only (about 2 cm long)
  Other Names: percutaneous compression-plate
  Arms: PCCP, Proximal femur fracture
Procedure: DHS — Conventional surgical treatment of proximal femur fracture including one longer approach from lateral
  Other Names: Dynamic hip screw
  Arms: DHS, proximal femur fracture
Procedure: Osteosynthesis with nails — Osteosynthesis with nails is a minimal-invasive surgery technique for proximal femur fractures.
  Arms: Osteosythesis with nails, prox. femur frac.

SUMMARY:
This project investigate any difference in inflammatory response,wound heeling rate, functional outcome and level of pain in patience with different surgical treatment (PCCT vs. DHS vs. Osteosynthesis with nails) after a fracture of the proximal femur.

DETAILED DESCRIPTION:
This project investigates microcirculation in skin and muscle after different surgical treatment of pertrochanteric fractures of the femur for detecting the less damaging method. Three different systems are compared: the PCCT and the osteosynthesis with nails ( two minimal-invasive methods) and the conventional dynamic hip screw ( DHS). All three are long established and show no difference in results in any clinical trials. The method for every patient is chosen randomly.

The microcirculation is measured as parameter for tissue damage and wound heeling. It is registered by O2c, which works with measuring reflected lightwaves. It is strictly noninvasive and causes absolutely no pain for the patient. The measurement device consists of two small probes, which simply stick to the patient´s skin. There are eleven measurements on this study: one directly before and one shortly after and one 6 h after the surgery, followed by three measuring appointments after 12, 24, 48 hours. Afterwards there are appointments planed after 4, 7 and 12 days. After 7 days a CT controls the leg-rotation. In addition it detects any dislocation of the fracture or fixing item.The next appointments are planed after 6 week. In the last two sessions the patients are questioned according to established questionnaires, e.g the Harris hip score to evaluate any loss of functionality of the operated leg. And a control of physical strength is planed on these appointments. It is known today that most patients can not reach the same level of physical strength after the treatment as before the fracture. Additionally an EMG records muscle damage. And the level of pain is evaluated with the Visual Analogue Scale simultaneity with the O2c-measurements.

The last measurement is planed after 6 month. Then the fracture is controlled by an X-ray.

Clinical parameters like operation time, blood loss, ASA score (for pre-existing condition) are included to create comparable patient profiles. Therefore the AO classification of the fracture and the grade of osteoporosis according to the Singh-Classification is recorded, too.

Also on every measuring appointment blood samples are tested on parameters of systemic inflammatory response and muscle cell destruction.

Furthermore this project is meant to establish limits of microcirculation measured with O2c. So in the future is will be possible to predict any wound heeling difficulties with this no-invasive measuring technic.

Therefore this study will research on the one hand if these three operation methods differ in wound heeling, functionality or level of pain and on the other hand establish a possibility to detect wound heeling complications early and easily.

Both results are extremely relevant to be able to choose the treatment most suited to the individual patient. So the pertrochanteric fracture of the femur, which is common in older and multimorbid population, will no longer result in risky re-operations due to wound heeling complications or limited functionality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Above 60 years of age
* Letter of approval firmed
* Proximal femur fracture

Exclusion Criteria:

* Pathologic fracture
* History of metabolic bone disease
* Earlier surgery s of the hip or femur on the same leg
* Fractures with osteosynthesis material of earlier treatment still in place
* Soft tissue damage
* Delay of surgery for more than 3 days
* Immune default
* Polytrauma
* Fracture ends more than 5 cm distal of trochanter minor

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Microcirculation | within 12 days
  The microcirculation is measured on different times by O2c to observe the trauma of surgery on skin and tissue and any wound healing difficulties.

SECONDARY OUTCOMES:
Systemic inflammatory response | within 12 days
  The systemic inflammatory response is monitored by different inflammatory parameters in blood samples, which are taken on several occasions post-op

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Pape, Univ-prof.MD, Study Chair — Chief of medicine
Locations (1):
- Universal Hospital of the RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany